CLINICAL TRIAL: NCT03959033
Title: A Pilot Study of Patient Reported Outcomes When Treated With Trabectedin for Unresectable and/or Metastatic Soft Tissue Sarcoma
Brief Title: Patient Reported Outcome Measures (PROMs) With Trabectedin
Status: Terminated | Type: Observational
Why Stopped: Insufficient accrual
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Daniel Stark, Associate Professor of Cancer Medicine, University of Leeds
Other Study IDs: 16/WM/0446
Record Dates: First submitted 2018-01-12; First posted 2019-05-22 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Sarcoma; Liposarcoma; Leiomyosarcoma
Keywords: PROMs; EORTC QLQc-30
MeSH Terms: conditions — Sarcoma; Liposarcoma; Leiomyosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patient reported outcome measures (PROMs) are central to understanding the impact of cancer treatments on patients. Treatment may control cancer growth, and even sometimes modestly improve the length of life, but at the expense of disruption of lifestyle, and of toxicities. It is very important to use PROMs to evaluate the balance between these risks and benefits to understand the overall impact of the treatment.

It remains poorly described whether patients report improved outcomes during palliative chemotherapy with trabectedin, using high quality questionnaires, and how this may vary with the clinical effects and duration of the treatment and characteristics of the patient.

DETAILED DESCRIPTION:
Trabectedin improves progression-free survival in un-resectable advanced soft tissue sarcoma, in particular lipo- and leiomyo- sarcomas after failure of conventional chemotherapy, with a low level of reported grade 3 symptomatic toxicity for many patients. However objective responses are infrequent, with the largest proportion of patients who benefit using traditional oncological response criteria having a delay in progression with the cancer stable. Trabectedin may improve the duration of cancer control by the modulation of cancer growth as measured by the growth modulation index (GMI).

Patient reported outcome measures (PROMs) are central to understanding the impact of cancer therapies which may shrink cancers or control their growth, and even sometimes modestly improve the length of life, but at the expense of disruption of lifestyle, and of toxicities.

It is very important to use PROMs to evaluate the balance between these risks and benefits to understand the overall impact of the therapy. It remains poorly described whether patients report improved outcomes during palliative chemotherapy with trabectedin, using validated questionnaires, and how this may vary with the clinical efficacy and duration of the treatment and the demographic and clinical characteristics of the patient. Therefore the investigators intend to examine the feasibility of collecting patient reported outcome measures using validated instruments prospectively during English NHS administration of Trabectedin and with this to explore the pattern of patient reported outcomes, such as is the trajectory in PROMs distinct comparing groups by the size or symptoms from tumour masses.

The study will aim deliver Patient Reported Outcomes Measures (PROMs) data in patients with advanced tissue sarcoma. The recruitment target is a total of 30 patients over a 2 year period. Patients' quality of life (QoL) will be captured using a validated QoL questionnaire (EORTC QLQ-C30) during their treatment with Trabectedin. The questionnaire takes approximately 12 minutes and the patient will complete this unaided. Patients will be required to complete the electronic questionnaire using Q-Tool. Q-Tool is a web-based piece of software. Patients will be required to complete this questionnaire alongside receiving standard of care treatment with Trabectedin in the following pattern: On the day of administration of the 1st of treatment with Trabectedin; before the 2nd treatment of Trabectedin; before the 4th treatment of Trabectedin; prior to the 7th treatment of Trabectedin; prior to the 10th treatment of Trabectedin and then will continue in 3 weekly cycles until the end of treatment with Trabectedin. Patients will complete the questionnaire on the computer terminals available in the outpatient clinic before they see the doctor and nurses and prior to treatment on each of these days.

Patients at the end of treatment with Trabectedin will complete a short exit questionnaire. This will assess their experiences of completing the QoL questionnaire and ease of using Q-Tool. The exit questionnaire will take approximately 5 minutes to complete. This will be completed in the outpatient area and provided to the patient by the Research Nurse.

ELIGIBILITY:
Inclusion Criteria:

* This study will include adult patients treated in Leeds with an indication for Trabectedin as either second or third line therapy for relapsed soft tissue sarcoma.
* Patients will have the ability to provide informed consent and they will have adequate literacy in reading English, or complete the instrument using an NHS interpreter.

Exclusion Criteria:

* No exclusion criteria

Ages: 16 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will identify adult patients treated in Leeds with an indication for Trabectedin as either second or third line therapy for relapsed soft tissue sarcoma.
  Patients suitable for treatment will be those with the following histologies Synovial Sarcoma Myxoid liposarcomas De-differentiated liposarcoma with some clinical sensitivity demonstrated to earlier lines of chemotherapy Leiomyosarcoma Other soft-tissue sarcomas with some clinical sensitivity demonstrated to earlier lines of chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Change in Global quality of life using the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire core 30 from baseline (week 1) through to 12 weeks (to day 1 of cycle 4 of trabectedin). | Through to study completion, an average of 12 weeks
  As this is a pilot exploratory study the investigators will have multiple co-primary outcomes.The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) is a 30 question assessment of quality of life in the following categories: global health status, physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning, fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea, and financial difficulties. Twenty-eight questions are assessed on a scale of 1 (Not at all) to 4 (Very much); 2 questions are assessed on a scale of 1 (very poor) to 7 (excellent). The range of scores on each scale is from 0 to 100. In the function scales, a score of 100 is best (indicating more function). In the symptom scores, a score of 100 is worst, indicating more symptoms. Scores are totalled from each item to form the scales, then normalised to 0-100.
What is the trajectory in the subscales and symptom scales in the scale, from baseline (day 1 cycle 1) to day 1 cycle 4, day 1 cycle 7 and day 1 cycle 10 etc of Trabectedin? | Through to study completion, an average of 12 weeks
  As this is a pilot exploratory study the investigators will have multiple co-primary outcomes.The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) is a 30 question assessment of quality of life in the following categories: global health status, physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning, fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea, and financial difficulties. Twenty-eight questions are assessed on a scale of 1 (Not at all) to 4 (Very much); 2 questions are assessed on a scale of 1 (very poor) to 7 (excellent). The range of scores on each scale is from 0 to 100. In the function scales, a score of 100 is best (indicating more function). In the symptom scores, a score of 100 is worst, indicating more symptoms. Scores are totalled from each item to form the scales, then normalised to 0-100.
What is the association between patient's prior treatment (second line versus third line) and the trajectory of the subscales and symptom scales in the EORTC QLQc30 ? | Through to study completion, an average of 12 weeks
  As this is a pilot exploratory study the investigators will have multiple co-primary outcomes.The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) is a 30 question assessment of quality of life in the following categories: global health status, physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning, fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea, and financial difficulties. Twenty-eight questions are assessed on a scale of 1 (Not at all) to 4 (Very much); 2 questions are assessed on a scale of 1 (very poor) to 7 (excellent). The range of scores on each scale is from 0 to 100. In the function scales, a score of 100 is best (indicating more function). In the symptom scores, a score of 100 is worst, indicating more symptoms. Scores are totalled from each item to form the scales, then normalised to 0-100.
What is the association between patient age (in deciles) and the trajectory of the subscales and symptom scales in the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire core 30 scale? | Through to study completion, an average of 12 weeks
  As this is a pilot exploratory study the investigators will have multiple co-primary outcomes.The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) is a 30 question assessment of quality of life in the following categories: global health status, physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning, fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea, and financial difficulties. Twenty-eight questions are assessed on a scale of 1 (Not at all) to 4 (Very much); 2 questions are assessed on a scale of 1 (very poor) to 7 (excellent). The range of scores on each scale is from 0 to 100. In the function scales, a score of 100 is best (indicating more function). In the symptom scores, a score of 100 is worst, indicating more symptoms. Scores are totalled from each item to form the scales, then normalised to 0-100.
What is the relationship between the trajectory of responses in the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire core 30 scale and the growth modulation index? | Through to study completion, an average of 12 weeks
  As this is a pilot exploratory study the investigators will have multiple co-primary outcomes.The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) is a 30 question assessment of quality of life in the following categories: global health status, physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning, fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea, and financial difficulties. Twenty-eight questions are assessed on a scale of 1 (Not at all) to 4 (Very much); 2 questions are assessed on a scale of 1 (very poor) to 7 (excellent). The range of scores on each scale is from 0 to 100. In the function scales, a score of 100 is best (indicating more function). In the symptom scores, a score of 100 is worst, indicating more symptoms. Scores are totalled from each item to form the scales, then normalised to 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Stark, Principal Investigator — University of Leeds; Daniel Stark, Principal Investigator — d.p.stark@leeds.ac.uk
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No